CLINICAL TRIAL: NCT03021291
Title: An Open-label Study Assessing the Effect of Gelesis100 on Weight Loss and Weight Maintenance in Overweight and Obese Subjects Who Completed the GLOW Study (G-04)
Brief Title: Extension Study of Gelesis100 on Body Weight
Acronym: GLOW-EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gelesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-100-009
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Gelesis100 (Experimental): Gelesis100 (2.25 g) twice daily
  Interventions: Device: Gelesis100 (2.25 g)

INTERVENTIONS:
Device: Gelesis100 (2.25 g) — Three capsules of Gelesis100, each containing a 750 mg mixture of two food-grade materials: carboxymethylcellulose that is cross-linked with citric acid.

SUMMARY:
This study is designed to assess the effect of Gelesis100 on body weight after an additional exposure of 24 weeks in subjects who completed the 24-week treatment period, and had at least 3% weight loss, in the Gelesis Loss Of Weight GLOW, NCT02307279) study.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of the GLOW study with at least 3% weight loss
2. Informed Consent Form signed by the subjects at the end of the GLOW study

Exclusion Criteria:

1. Pregnancy (or positive serum or urine pregnancy test(s) in females of childbearing potential) or lactation
2. Absence of medically approved contraceptive methods in females of childbearing potential (e.g., hysterectomy, non-oral contraceptive medications or intrauterine device combined with a barrier method, two combined barrier methods such as diaphragm and condom or spermicide, or condom and spermicide; bilateral tubal ligation and vasectomy are not acceptable contraceptive methods)
3. Subjects considering smoking cessation during the study
4. Subjects anticipating surgical intervention during the study
5. Significant intolerance to the study product during the GLOW study
6. Increase of ≥ 0.5% point (≥ 5.5 mmol/mol) in HbA1c from the Baseline Visit of the GLOW study in subjects with treated or untreated type 2 diabetes if considered clinically relevant, or any increase if HbA1c is > 8.5% (> 69 mmol/mol)
7. Increase of ≥ 10% in total cholesterol, low-density lipoprotein (LDL) cholesterol, or triglycerides from the Baseline Visit of the GLOW study in subjects with elevated lipids at the Baseline Visit of the GLOW study if considered clinically relevant, or any increase if serum LDL cholesterol is ≥ 190 mg/dL (≥ 4.93 mmol/L) and/or serum triglycerides are ≥ 500 mg/dL (≥ 5.65 mmol/L)
8. Increase of ≥ 10 mm Hg in supine systolic blood pressure (SBP) and/or supine diastolic blood pressure (DBP) from the Baseline Visit of the GLOW study in subjects with treated or untreated hypertension if considered clinically relevant, or any increase if supine SBP is > 160 mm Hg and/or supine DBP is > 95 mm Hg, based on the mean of two consecutive readings
9. Poor subject compliance with the GLOW study procedures and recommendations and/or major protocol deviation
10. Anticipated requirement for use of prohibited concomitant medications

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Percent (%) change from baseline
Body weight responders (5%) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in body weight of at least 5%

SECONDARY OUTCOMES:
Change in plasma glucose status (normal, impaired, diabetic) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
Change in plasma glucose | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in millimoles per liter (mmol/L)
Change in insulin resistance | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in homeostatic model assessment of insulin resistance (HOMA-IR)
Change in glycosylated hemoglobin (HbA1c) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (%)
Change in body mass index (BMI) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Measured as body weight in kilograms divided by height in meters-squared (kg/m2)

OTHER OUTCOMES:
Body weight responders (10%) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in body weight of at least 10%
Change in excess body weight | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (%)
Change in body weight status (normal, overweight, obese) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
Change in waist circumference | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in waist circumference (centimeters)
Change in serum insulin | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in milliunits per liter (mU/L)
Change in serum C-reactive protein (CRP) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Measured in milligrams per liter (mg/L)
Change in total cholesterol, serum low-density lipoprotein (LDL), high-density lipoprotein (HDL), total cholesterol/HDL ratio, and triglycerides | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  measured in milligrams per deciliter (mg/dL)
Change vital signs: heart rate, supine and standing systolic and diastolic blood pressure (SBP, DBP) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Measured in beats per minute (heart rate) or millimeters of mercury (mmHg) for blood pressure
Change in food intake | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Assessed by 24 hr dietary recall
Change in Impact of Weight on Quality Of Life (IWQOL) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change in global and individual questionnaire subscale scores
All adverse events (AE), serious adverse events (SAE), and gastrointestinal symptoms | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Number and % of subjects with AE/SAEs spontaneously reported; gastrointestinal symptoms solicited via questionnaire.
Change in serum sodium | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in millimoles per liter (mmol/L)
Change in serum potassium | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (mmol/L)
Change in serum chloride | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (mmol/L)
Change in serum calcium | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (mmol/L)
Change in serum magnesium | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (mmol/L)
Change in serum phosphorus | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (mmol/L)
Change in serum glucose | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (mmol/L)
Change in blood urea nitrogen (BUN) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (mmol/L)
Change in serum creatinine | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in micromoles per liter (umol/L)
Change in serum uric acid | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (umol/L)
Change in total bilirubin | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (umol/L)
Change in alanine aminotransferase (ALT) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline in international units per liter (IU/L)
Change in aspartate transaminase (AST) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (IU/L)
Change in gamma-glutamyl transpeptidase (GGT) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (IU/L)
Change in alkaline phosphatase (ALP) | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (IU/L)
Change in serum total protein | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (g/L)
Change in serum albumin | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (g/L)
Change in hematocrit | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (%)
Change in hemoglobin | Measured at baselines of the GLOW and GLOW-EX study (day 197) and day 339
  Change from baseline (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Heshmati, MD, Study Director — Gelesis, Inc.
Locations (16):
- United States (11):
  - Arternis Institute for Clinical Research, San Diego, California
  - Clinical Trial Investigators, Tustin, California
  - University of Colorado, Aurora, Colorado
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Pennington Biomedical Research, Baton Rouge, Louisiana
  - Boston University Medical Center, Boston, Massachusetts
  - Cornell Weill Medical College, New York, New York
  - Radiant Research, Cincinnati, Ohio
  - Aventiv Research, Columbus, Ohio
  - Geisinger Health System, Danville, Pennsylvania
  - Texas Diabetes and Endocrinology, Round Rock, Texas
- Health & Care SRO, Prague, Czechia
- University of Cophenhagen, Copenhagen, Denmark
- Italy (2):
  - IRCCS Policlinico San Donato, Milan
  - University of Rome, Rome
- University of Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: Undecided